CLINICAL TRIAL: NCT06444204
Title: An Open-Label, Phase 1 Study to Evaluate the Effect of Mild and Moderate Hepatic Impairment on the Single-Dose Pharmacokinetics of Rilzabrutinib (PRN1008)
Brief Title: A Study to Evaluate the Effect of Mild and Moderate Hepatic Impairment on the Single-Dose Pharmacokinetics of Rilzabrutinib (PRN1008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP17091; U1111-1260-4098 (Registry Identifier: ICTRP); PRN1008-020 (Other: Sanofi Identifier); POP17091 (Other: Sanofi Identifier)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Hepatic Function Abnormal; Healthy Volunteers
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rilzabrutinib: Mild Hepatic Impairment (Experimental): Subjects with mild Hepatic Impairment (HI)
  Interventions: Drug: Rilzabrutinib
- Rilzabrutinib: Moderate Hepatic Impairment (Experimental): Subjects with moderate Hepatic Impairment (HI)
  Interventions: Drug: Rilzabrutinib
- Rilzabrutinib: Healthy-Matched Control (Experimental): Subjects with normal hepatic function
  Interventions: Drug: Rilzabrutinib

INTERVENTIONS:
Drug: Rilzabrutinib — Rilzabrutinib tablet administered orally

SUMMARY:
This is a single-dose study to assess the effect of mild or moderate Hepatic Impairment (HI) on the Pharmacokinetics (PK) of rilzabrutinib as well as to evaluate the safety and tolerability of rilzabrutinib in subjects with HI.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic Impaired Subjects:

  * Non-smoking or light smoker (not exceeding 5 cigarettes per day), adult male or non-pregnant, non-lactating female, 18-75 years of age, inclusive, at screening.
  * Weight ≥ 50 kg, at screening.
* Healthy Subjects:

  * Non-smoking or light smoker (not exceeding 5 cigarettes per day), healthy, adult males and non-pregnant, non-lactating females, 18-75 years of age, inclusive, at screening.

Subject must be matched for age (within ± 10 years), and sex of the matched subject with hepatic impairment.

--Weight ≥ 50 kg at screening.

Additional inclusion criteria might apply.

Exclusion Criteria:

* Hepatic Impaired Subjects:

  * Pregnant or lactating female.
  * Uncontrolled treated/untreated hypertension (systolic blood pressure ≥ 160 millimeters of mercury [mmHg] and/or diastolic blood pressure ≥ 105 mmHg), or resting pulse rate < 45 or > 100 beats per minute (bpm). Measurements may be repeated once in order to determine eligibility.
* Healthy Subjects

  * Pregnant or lactating female.
  * Uncontrolled treated/untreated hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 105 mmHg), or resting pulse rate < 45 or > 100 bpm. Measurements may be repeated once in order to determine eligibility.

Additional exclusion criteria might apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of total rilzabrutinib in plasma from 0 to t (AUC0-t) | Up to 30 hours after rilzabrutinib dosing
Area under the concentration-time curve of total rilzabrutinib in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | Up to 30 hours after rilzabrutinib dosing
Percent of AUC0-inf extrapolated total rilzabrutinib in plasma (%AUCextrap ) | Up to 30 hours after rilzabrutinib dosing
Maximum measured concentration of total rilzabrutinib in plasma (Cmax) | Up to 30 hours after rilzabrutinib dosing
Time from dosing to maximum measured concentration of total rilzabrutinib in plasma (tmax) | Up to 30 hours after rilzabrutinib dosing
Terminal Half-Life of total rilzabrutinib in Plasma (t1/2) | Up to 30 hours after rilzabrutinib dosing
Elimination Rate Constant of total rilzabrutinib (Kel) | Up to 30 hours after rilzabrutinib dosing
Apparent Total Clearance of rilzabrutinib in the plasma after extra-vascular administration (CL/F) | Up to 30 hours after rilzabrutinib dosing
Apparent Volume of Distribution during the Terminal elimination phase after extravascular administration (Vz/F) | Up to 30 hours after rilzabrutinib dosing
Fraction of unbound drug ( rilzabrutinib) expressed as percent (%fu) | Up to 24 hours after rilzabrutinib dosing
Number of Adverse Events (AE) / Serious Adverse Events (SAE) | From date of signed ICF, up to 9 days after rilzabrutinib dosing
Incidence of potentially clinically significant laboratory test, vital signs, and electrocardiogram (ECGs) abnormalities | Up to 30 hours after rilzabrutinib dosing

SECONDARY OUTCOMES:
Area under the concentration-time curve of rilzabrutinib metabolites in plasma from 0 to t (AUC0-t) | Up to 24 hours after rilzabrutinib dosing
Area under the concentration-time curve of rilzabrutinib metabolites in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | Up to 24 hours after rilzabrutinib dosing
Percent of AUC0-inf extrapolated rilzabrutinib metabolites in plasma (%AUCextrap) | Up to 24 hours after rilzabrutinib dosing
Maximum measured concentration of rilzabrutinib metabolites in plasma (Cmax) | Up to 24 hours after rilzabrutinib dosing
Time from dosing to maximum measured concentration of rilzabrutinib metabolites in plasma (tmax) | Up to 24 hours after rilzabrutinib dosing
Terminal Half-Life of rilzabrutinib metabolites in Plasma (t1/2) | Up to 24 hours after rilzabrutinib dosing
Elimination Rate Constant of rilzabrutinib metabolites (Kel) | Up to 24 hours after rilzabrutinib dosing
Metabolite-to-parent ratio (MRAUC) | Up to 24 hours after rilzabrutinib dosing
  MRAUC is Based on AUC0-t, corrected for Molecular weights (MW). MRAUC = (AUC0-t,M/AUC0-t,P) x (MW,P/MW,M) where M was metabolite and P was parent.
Metabolite-to-parent ratio (MRCmax) | Up to 24 hours after rilzabrutinib dosing
  MRCmax is based on Cmax, corrected for MW. MRCmax = (Cmax,M/ Cmax,P) x (MW,P/MW,M) where M was metabolite and P was parent.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Investigational Site Number: 0002, Miami, Florida
  - Investigational Site Number: 0001, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org